CLINICAL TRIAL: NCT02628509
Title: Onset and Offset of Von Willebrand Factor Multimemirization Defects in Cardiovascular Disease: the Case of the Molecular Sensor of Blood Flow
Brief Title: Von Willebrand Factor As a Biological Sensor of Blood Flow in Percutaneous Cardiac Procedure
Acronym: WiTAVi
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: NI_59
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Heart Failure; Aortic Stenosis
Keywords: Acquired Von Willebrand; Trans aortic valve replacement; mechanical circulatory support
MeSH Terms: conditions — Heart Failure; Aortic Valve Stenosis | interventions — Cardiac Resynchronization Therapy Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiac devices: patients receiving mechanical circulatory support patients undergoing transaortic valve replacement
  Interventions: Device: cardiac devices

INTERVENTIONS:
Device: cardiac devices — patients receiving mechanical circulatory support or undergoing trans aortic valve replacement
  Other Names: trans aortic valve replacement; mechanical circulatory support

SUMMARY:
The WITAVI study was designed to explore the kinetic and associated outcome of Von Willebrand Factor-multimerizaton defects associated with devices in cardiovascular diseases.

DETAILED DESCRIPTION:
This study was designed to understand the Von Willebrand Factor (VWF) abnormalities observed in association with implantation of different devices in cardiovascular diseases (percutaneous valve replacement and circulatory support devices).

The main objective of the study was to describe the time-course of VWF abnormalities onset/offset during implantation of devices in cardiovascular diseases.

Adult patients > 18 years who need a CF-LVAD or trans-aortic valve implantation are included in this cohort; Blood samples are obtained just before procedures

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years who need a mechanical circulatory support due to advanced heart failure or undergoing trans-aortic-valve-replacement to treat aortic stenosis.
* Informed consent of the patient or support person in case of disability at baseline (patient intubated and ventilated)

Exclusion Criteria:

* Patient with a known severe bleeding disorder
* Patient refusal or environment
* Minor patients
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients receiving mechanical circulatory support or undergoing aortic valve replacement
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-08 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Von Willebrand factor (VWF) multimer defects | 180 minutes after device implantation
  VWF multimeric analysis is performed by electrophoresis. The results of HMW-multimers are expressed as the relative amount of the largest multimers (mer>15) of the sample compared with those of the normal pooled plasma (NPP standard human plasma Siemens healthcare diagnostics, Marburg, Germany, coefficient of variation=11%) present on each gel. 4-6 With this method the HMW-multimer ratio is defined as the HMW-multimers (>15-mer) in patient plasma sample divided by HMW-multimers in normal pool plasma, the HMW-multimer ratio of normal pooled plasma is 1 (by definition) and an HMW-multimer defect is defined as a reduced HMW-multimer-ratio (<1).

SECONDARY OUTCOMES:
platelet function analyser- ADP (PFA-ADP) closure time | 5, 15,30, 60 minutes; day 1 , day 7 after device implantation
  The PFA test is initially performed with the Collagen/Epinepherine membrane. A normal Col/ADP closure time (<180 seconds) excludes the presence of a significant platelet function defect.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Susen, MD, PhD, Study Chair — Lille University Hospital
Locations (1):
- Lille University Hospital, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Belle E, Rauch A, Vincentelli A, Jeanpierre E, Legendre P, Juthier F, Hurt C, Banfi C, Rousse N, Godier A, Caron C, Elkalioubie A, Corseaux D, Dupont A, Zawadzki C, Delhaye C, Mouquet F, Schurtz G, Deplanque D, Chinetti G, Staels B, Goudemand J, Jude B, Lenting PJ, Susen S. Von Willebrand factor as a biological sensor of blood flow to monitor percutaneous aortic valve interventions. Circ Res. 2015 Mar 27;116(7):1193-201. doi: 10.1161/CIRCRESAHA.116.305046. Epub 2015 Feb 10. PMID 25670067
- [Derived] Vincent F, Spillemaeker H, Kyheng M, Belin-Vincent C, Delhaye C, Pierache A, Denimal T, Verdier B, Debry N, Moussa M, Schurtz G, Porouchani S, Cosenza A, Juthier F, Pamart T, Richardson M, Coisne A, Hertault A, Sobocinski J, Modine T, Pontana F, Duhamel A, Labreuche J, Van Belle E. Ultrasound Guidance to Reduce Vascular and Bleeding Complications of Percutaneous Transfemoral Transcatheter Aortic Valve Replacement: A Propensity Score-Matched Comparison. J Am Heart Assoc. 2020 Mar 17;9(6):e014916. doi: 10.1161/JAHA.119.014916. Epub 2020 Mar 16. PMID 32172643
- [Derived] Van Belle E, Rauch A, Vincent F, Robin E, Kibler M, Labreuche J, Jeanpierre E, Levade M, Hurt C, Rousse N, Dally JB, Debry N, Dallongeville J, Vincentelli A, Delhaye C, Auffray JL, Juthier F, Schurtz G, Lemesle G, Caspar T, Morel O, Dumonteil N, Duhamel A, Paris C, Dupont-Prado A, Legendre P, Mouquet F, Marchant B, Hermoire S, Corseaux D, Moussa K, Manchuelle A, Bauchart JJ, Loobuyck V, Caron C, Zawadzki C, Leroy F, Bodart JC, Staels B, Goudemand J, Lenting PJ, Susen S. Von Willebrand Factor Multimers during Transcatheter Aortic-Valve Replacement. N Engl J Med. 2016 Jul 28;375(4):335-44. doi: 10.1056/NEJMoa1505643. PMID 27464202